CLINICAL TRIAL: NCT01922804
Title: Investigations of the Effect of MK-7 on Bone and Glucose Metabolism and Arterial Calcification
Acronym: K2vita
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Axellus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K2vita
Record Dates: First submitted 2013-08-06; First posted 2013-08-14 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Metabolic Bone Disorder
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- K2 vitamin (Experimental): K2 vitamin 375 microgram a day for 3 years
  Interventions: Dietary Supplement: K2 vitamin
- placebo (Placebo Comparator): 1 tablet a day for 3 years
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: K2 vitamin — K2 vitamin tablet
  Arms: K2 vitamin
Dietary Supplement: Placebo — Placebo tablets
  Arms: placebo

SUMMARY:
The aims of the present study are to investigate the effect of vitamin K2 on bone turnover, bone mass, bone structure, glucose metabolism, and arteriosclerosis.

Osteoporosis, diabetes, metabolic syndrome and cardiovascular disease are common diseases that affect large groups of people in the Western world.

Our hypotheses is that vitamin K2 (MK-7) reduces undercarboxylated osteocalcin in postmenopausal women and reduces bone turnover and increases bone mineral density; increases insulin sensitivity and decreases indices of arterial calcification.

DETAILED DESCRIPTION:
Osteoporosis, diabetes, metabolic syndrome and cardiovascular disease are common diseases that affect large groups of people in the Western world.

Our hypotheses is that vitamin K2 (MK-7) reduces undercarboxylated osteocalcin in postmenopausal women and reduces bone turnover and increases bone mineral density; increases insulin sensitivity and decreases indices of arterial calcification.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* 60-80 years
* osteopenia

Exclusion Criteria:

* Calcium metabolic, thyroid, liver or kidney disease
* Diabetes
* Obesity
* Myocardial infarction or other arteriosclerotic events
* Angina pectoris
* Vitamin D < 50 nmol/L
* Treatment with vitamin K antagonists
* Use of vitamin K supplements in the last month or for more than 3 months at any time
* Treatment with drugs with known effects on bone metabolism or glucose metabolism.
* Smoking in the last 12 months
* Drug or alcohol abuse
* Allergy to calcium, vitamin D or vitamin K.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
p-undercarboxylated osteocalcin | Change in undercarboxylated osteocalcin in plasma after 3 month treatment compared to baseline. Analysed in batch after the end of trial.

SECONDARY OUTCOMES:
Change in bone mineral density | Assessed after 3, 6, 12, 24 and 36 months
  Change in bone mineral density measured by DXA scans (Dual energy x-ray absorptiometry)
Change in arterial stiffness, pulse wave velocity | Measured at baseline and after 6 months
  Change in pulse wave velocity after 6 months.
Change in insulin sensitivity | Measured at baseline and after 1 and 12 months.
  Change in insulin sensitivity. Determined by HOMA-test (homeostasis model assessment), using fasting plasma glucose and insulin.
Change in bone turnover markers | Measured at baseline, after 1, 3, 6, 12, 24 and 36 months
Change in bone structure | baseline and month 12
  HRpQCT scans

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Rønn, cand.med, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Endocrinology and Internal Medicine THG, Aarhus, Denmark

REFERENCES:
- [Derived] Ronn SH, Harslof T, Oei L, Pedersen SB, Langdahl BL. The effect of vitamin MK-7 on bone mineral density and microarchitecture in postmenopausal women with osteopenia, a 3-year randomized, placebo-controlled clinical trial. Osteoporos Int. 2021 Jan;32(1):185-191. doi: 10.1007/s00198-020-05638-z. Epub 2020 Oct 8. PMID 33030563